CLINICAL TRIAL: NCT06312150
Title: Retro-prospective Observational Study on the Role of the β3 Adrenergic Receptor as a Tumour Biomarker in Paediatric Solid Tumours
Brief Title: Role of Tumoral Biomarker B3 Adrenergic Receptor in Paediatric Solid Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Annalisa Tondo, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BETA 3 2019
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with tumour (age 0-20 years) (Other): Patients affected by Wilms' tumour, Ewing's Sarcoma, Osteosarcoma, Soft tissue sarcomas, Carcinomas, Neuroblastoma age between 0-20 years
  Interventions: Other: Analysis of biological sample (Substudy-solid neoplasms)
- Patients with tumour (age 0-75 years) (Other): Patients affected by Ewing's Sarcoma, Neuroblastoma, Paediatric leukaemia, Breast, lung, colon and ovarian cancers between 0-75 years
  Interventions: Other: Analysis of biological sample (substudy-leukaemia patients)
- Control Patients group (Other): Patients underwent their diagnostic pathway, which made it possible to exclude the presence of any ongoing pathological process
  Interventions: Other: Analysis of peripheral blood (control group)

INTERVENTIONS:
Other: Analysis of peripheral blood (control group) — Peripheral blood sample will be acquired in excess to the last scheduled control sample according to clinical practice.
  Arms: Control Patients group
Other: Analysis of biological sample (Substudy-solid neoplasms) — peripheral blood sample, bone marrow aspirate and fresh or paraffin biopsia tissutale will be collected for the substudy
  Arms: Patients with tumour (age 0-20 years)
Other: Analysis of biological sample (substudy-leukaemia patients) — sample of peripheral blood and bone marrow blood for the substudy, derived from paediatric or young adult leukaemia patients
  Arms: Patients with tumour (age 0-75 years)

SUMMARY:
Childhood cancers are the third leading cause of death among children between the ages of 1 and 4, and the second leading cause of death among children aged 5-14 years. Biologically, it has been demonstrated that tumour aggressiveness and invasive capacity are caused by genetic modifications and cellular microenvironmental factors in a sequential and multifactorial process. The search for genetic alterations, proteins, or entire intracellular signalling pathways involved in the process of carcinogenesis and metastatisation is always evolving in order to identify new prognostic factors or potential therapeutic targets. In recent years, β-adrenergic receptors (β-ARs) have been associated with tumour progression.

This is a multicentre biological samples study which main aim is to evaluate the β3 receptor expression in the peripheral blood of patients with solid tumours compared to a healthy control group. The biological samples collected during the study are: peripheral blood sample, bone marrow aspirate and fresh or fresh paraffin biopsy tumour.

ELIGIBILITY:
Inclusion Criteria (principal study):

* Diagnoses, received after the year 2015 (Wilms' tumour, Ewing's Sarcoma, Osteosarcoma, Soft tissue sarcomas, Carcinomas, Neuroblastoma)
* Informed consent signed by parents or the patient if over 18 years of age
* Planned follow-up for 5 years
* Availability of a sufficient peripheral blood sample for analysis at onset.
* Age between 0 and 20 years

Inclusion Criteria (substudy):

* Diagnosis of Ewing's Sarcoma, Neuroblastoma, Paediatric leukaemia, Tumours of the breast, lung, colon and ovary
* Informed consent signed by parents or by the patient if 18 years of age19
* Planned follow-up for 5 years
* Availability of biological samples (peripheral blood, bone marrow blood, biopsy at onset) sufficient for the study investigations.
* Age between 0 and 20 years for paediatric patients referred to CROP Centres - Florence and Pisa
* Age between 19 and 75 years for adult patients attending the San Donato Hospital in Arezzo

Inclusion criteria (control group)

* Age between 0 and 30 years
* No evidence of acute or chronic infectious/inflammatory disease

Exclusion Criteria (for every partecipants to the principal study and substudy):

* Patients with HIV, HCV and HBV seropositivity (HBSAg) due to biohazard and bias related to patients' immunological status that could influence gene expression and tumour behaviour.
* Pregnant or lactating patients as the altered hormonal panel is a factor disturbing the expression of β3ARs

Ages: 1 Day to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of β3 receptor expression in the peripheral blood, bone marrow and bioptic samples of patients with solid tumours compared to a healthy control group | through study completion, an average of 1 year
  Cytofluorimetric data following labelling with specific fluorescent antibodies and after specific gating strategy, specific for each tumour or healthy cell, will be reported as a percentage (%), mean or median expression on the viable population of cells expressing the receptor. Data will be acquired at the MacsQuant Miltenyi Biotech cytofluorometer and analysed withFlowLogic® software programme.
Assessment of oxidative stress in peripheral blood samples from enrolled patients | through study completion, an average of 1 year
  Oxidative stress in the peripheral blood of patients enrolled in the main study will be assessed and healthy subjects, through the use of the Callegari instrument by measuring the amount of free radicals and antioxidants in the sample under analysis using specific detection kits.

SECONDARY OUTCOMES:
Evaluation of the role of the β3 receptor in apoptosis resistance (substudy) | through study completion, an average of 1 year
  Cells properly isolated and resuspended in PBS (phosphate buffered saline) will be incubated at room temperature with specific antibodies for Annessin V and Propidium Iodide (PI) compound and subsequently evaluated by flow cytometry (FACS).

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ospedale San Donato di Arezzo, Arezzo
  - Meyer Children's Hospital IRCCS, Florence
  - Azienda Ospedaliera Pisana, Pisa